CLINICAL TRIAL: NCT02545062
Title: Early Detection of Mild Cognitive Impairment in Young Diabetes Patients Using the MoCa Test
Brief Title: MoCa Test for the Early Detection of Mild Cognitive Impairment During Annual Assessment of Young Adults With Diabetes and in a Control Group Without Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Clalit Health Services (Other)
Responsible Party: Principal Investigator, Viviana Ostrovsky, Dr. (MD) (specialist in Internal Medicine and Endocrinology and Diabetes), Clalit Health Services
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DM- MOCA- 1
Record Dates: First submitted 2015-08-23; First posted 2015-09-09 (Estimated); Last update posted 2015-09-11 (Estimated); Status verified 2015-09

CONDITIONS: Diabetes Mellitus Type 1; Diabetes Mellitus Type 2; Mild Cognitive Impairment
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- group of type 1 and 2 diabetics (Experimental): A group of type 1 and 2 diabetes patients who meets the inclusion criteria will be done the MoCa test. A fingertip blood glucose will be made previous to the begin with the test in order to avoid doing it on a hypoglycemia event. The participants are instructed to do or respond the items in a organized manner. For each items there's a score. If the participant has 12 years of education or fewer, a point is added to his total score. At the end of the test the investigator will sum all sub items scores listed on the right side of the test paper. The maximum score is 30.
  The MoCa test will be done in a control group, no diabetics, that meets the inclusion criteria.
  Interventions: Other: MoCa test
- control group (Experimental): The MoCa test will be done in a control group, no diabetics, that meets the inclusion criteria.
  Interventions: Other: MoCa test

INTERVENTIONS:
Other: MoCa test — The MoCa test is actually used for the screening of Mild Cognitive Impairment . It is a one page 30 points test that can be done in 10 minutes in a routine annual visit to the Diabetes Clinic. The MoCa assesses several cognitive domains, and it is available in hebrew language.

SUMMARY:
T2D and cognitive impairment are two of the most common chronic condition found in persons 60 years and older. Diabetes type 2 increases with age and studies suggest that the diabetes is one of the risk factor for cognitive impairment and dementia.

Although there is much recent research showing that diabetics at every age have more cognitive impairment and dementia than non-diabetics, relatively little attention has been paid to the implications of this complication in the management of T2D in terms of screening, prevention, education and treatment adherence.

There are now guidelines for periodic evaluation of patients with diabetes as early detection of complications of the disease, but so far there are no similar assessment and monitoring of cognitive function.

In this study the investigators examine cognitive function in young diabetic patients (from 20 to 55) using the MoCa test, that allows detection of mild cognitive impairment, and may be carried out during a visit, an annual advisory diabetes clinic.

DETAILED DESCRIPTION:
1. Patients on a routine visit to the diabetes clinic, who meet the inclusion criteria, will be recruited for the test. They will be given an explanation of the study and the questionnaire by the principal investigator.
2. Sign a consent form.
3. Performance and execution of MOCA test:

   * Fingerstick blood glucose for pre-cognitive testing performed (to avoid testing any participant with a serum glucose < 70 mg/dl);
   * In the presence of hypoglycemia, the participant should be given a snack and begin the test only after the glucose level rises. Alternatively delay executing the Test
4. Details from the patient's file are registered, such as: duration of the disease, family history, presence of macro and micro vascular complications, lifestyle, years of education, and the results of relevant laboratory accuracy.
5. For each patient a medical file is opened containing the initials and serial number of his research. All results are then encoded and analyzed anonymously

ELIGIBILITY:
Inclusion Criteria:

* type 1 and 2 diabetes meIlitus
* 20 to 55 years old
* up to 15 years of diabetes disease duration
* fluent speech and read hebrew's language only

Exclusion Criteria:

* not meeting the inclusion criteria
* psychiatric disease
* dementia
* chronic use of alcohol or illegal drugs
* use of medication that can alter the attention or cognition of the participant
* active cardiovascular disease in the previous six months before the investigation
* oncology disease in the previous six months before the investigation

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 170 (Estimated)
Dates: Start 2014-05; Primary Completion 2016-08 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
The differences between the MoCa test score in diabetics and in a control group of non diabetics | 1 year

SECONDARY OUTCOMES:
The relation between the MoCa test score and glycemic control, in terms of HA1C value, in the past year before recruitment | 1 year
The relation between the MoCa test score and the presence of microvascular complications, retinopathy, polyneuropathy and nephropathy | 1 year
The relation between the MoCa test score and the presence of macrovascular complication, ischemic heart disease, non-fatal myocardial infarct, stable and unstable angina, heart failure, non-fatal stroke, peripheral vascular disease | 1year

CONTACTS AND LOCATIONS:
Overall Officials: Joel JS Singer, MD, Study Director — Clalit Medical Service
Locations (1):
- Viviana Ostrovsky, Nes Tziona, Israel, Israel